CLINICAL TRIAL: NCT07180147
Title: Arlington Longitudinal Optimal Healthy Aging Study (ALOHA)
Acronym: ALOHA
Status: Recruiting | Type: Observational
Sponsor: Marymount University (Other)
Collaborators: Potomac Health Foundations (Other)
Responsible Party: Principal Investigator, Patricia C. Heyn, Vice President for Research, Marymount University
Other Study IDs: MUIRB#1238; Potomac Health Foundation (Other Grant/Funding Number: 2025-2026 Howard L. Greenhouse Grant)
Record Dates: First submitted 2025-08-15; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease (AD); Cardio Vascular Disease; Mild Cognitive Impairment (MCI); Frailty Syndrome; Disability Physical; Hypertension; Metabolic Syndrome (MetS); Healthy Aging; Obesity &Amp; Overweight
Keywords: Optimal aging; dementia risk factors; Cardiovascular Health; Healthy Aging; Alzheimer Disease Prevention; Lifestyle Intervention; Dementia Risk Reduction; Cognitive Aging; Brain Health; Falls Prevention; Physical Function; Functional Independence; Frailty Prevention; Modifiable Risk Facators
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Frailty; Hypertension; Metabolic Syndrome; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALOHA Health Passport Cohort: Community-dwelling adults aged 50 and older who receive a comprehensive baseline and annual health assessment at the Marymount University Center for Optimal Aging. Assessments include physical, cognitive, and psychosocial measures. Results are compiled into a personalized "Health Passport" with tailored recommendations for managing modifiable health risk factors. Participants return annually for up to 5 years to monitor health changes, update recommendations, and complete follow-up surveys on adherence and outcomes.

SUMMARY:
The Arlington Longitudinal Optimal Healthy Aging (ALOHA) Study is a community-based research project led by the Marymount University Center for Optimal Aging (MCOA). The study is designed to help older adults in the Washington, D.C., Maryland, and Virginia (DMV) area maintain independence, mobility, wellbeing and brain health as they age.

Adults aged 50 years and older will receive a comprehensive health assessment at the study site, Center for Optimal Aging- ALOHA Lab at Marymount University (MU) Ballston Campus in Arlington, Virginia. The assessment includes physical and cognitive testing, health and medical history, lifestyle surveys, and biometric measures such as blood pressure, grip strength, body composition by the InBody system, balance and gait speed. Participants will receive their results in a personalized "Health Passport," which summarizes findings and provides tailored recommendations to help manage modifiable health risk factors-such as those linked to Alzheimer's disease, cardiovascular disease, frailty syndrome, and depression.

Participants will return annually for up to 5 years to repeat assessments and receive updated health and wellness recommendations. The study will track changes in health over time and explore the impact of the Health Passport on health behaviors, functional independence, and quality of life. ALOHA will also evaluate the cultural appropriateness of the Health Passport for diverse populations in Northern Virginia.

The program incorporates an interprofessional research model, engaging researchers from multiple health professions to work alongside older adults, supporting both participants' wellness and optimal aging.

DETAILED DESCRIPTION:
The Arlington Longitudinal Optimal Healthy Aging (ALOHA) Study is an interdisciplinary, mixed-method, longitudinal research program aimed at identifying, tracking, and managing modifiable health risk factors that influence optimal aging. The study serves community-dwelling adults aged 50 and older living in the DMV region, with initial recruitment focused on healthy individuals without significant cognitive impairment or terminal illness.

The ALOHA framework combines comprehensive baseline and follow-up health assessments with personalized wellness guidance. At enrollment, participants undergo:

1. Physical health evaluations (vital signs, body composition via bioimpedance, cardiovascular function via arteriography, mobility and endurance tests, grip strength, flexibility, balance)
2. Cognitive assessments (Montreal Cognitive Assessment, Central Nervous System [CNS] Vital Signs, Wechsler Memory and Intelligence scales, Quality of Life in Neurological Disorders [Neuro-QOL] Cognitive Function survey)
3. Lifestyle and psychosocial surveys (physical activity, diet quality using the MIND diet score, depression screening via the Center for Epidemiologic Studies Depression Scale [CES-D], social determinants of health, oral health, self-efficacy, quality of life)

Findings are compiled into a tailored, participant-specific, "Health Passport," which summarizes results in accessible language and offers practical, evidence-based recommendations for reducing disease risk, improving physical and cognitive function, and promoting overall wellness.

Participants return annually for up to five years to repeat assessments, receive an updated Health Passport consultation, and complete follow-up surveys regarding adherence, satisfaction, and changes in health status. The longitudinal design allows researchers to examine health trajectories, the effectiveness of early prevention strategies, and the relationship between modifiable risk factors and outcomes such as functional independence and cognitive decline.

Primary study aims:

1. Identify and track the prevalence of modifiable risk factors for Alzheimer's disease, cardiovascular disease, frailty, and depression.
2. Provide tailored recommendations to support participant-driven health improvement and evaluate adherence to Health Passport guidance.
3. Engage older adults and university students in an intergenerational, interprofessional health promotion research model.

The study emphasizes cultural inclusivity, particularly for Northern Virginia's racially and ethnically diverse populations. Spanish-language materials and validated translated assessments are incorporated to support Hispanic/Latino participants.

By integrating clinical, behavioral, and community health approaches, the ALOHA study aims to contribute new evidence on preventive aging strategies, refine the Health Passport model, and expand its use to other communities and academic centers.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older at time of enrollment
* Residing in the Washington, District of Columbia (DC)., Maryland, or Virginia metropolitan areas
* Community-dwelling (living independently or with minimal assistance)
* Able to participate in physical and cognitive assessments
* Able to provide informed consent
* Willing to return for annual follow-up assessments for up to 5 years

Exclusion Criteria:

* Diagnosis of dementia or significant cognitive impairment that prevents informed consent or participation in assessments
* Severe physical disability or medical condition that precludes participation in study assessments (e.g., unstable cardiac condition, severe mobility limitation)
* Current diagnosis of a terminal illness with life expectancy less than 12 months
* Residing in a long-term care facility or nursing home at time of enrollment
* Inability to communicate in English or Spanish (study materials available in these languages only)
* Participation in another interventional trial that could confound study results

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults aged 50 years and older living in the Washington, D.C., Maryland, and Virginia metropolitan area. Participants are generally healthy or have manageable chronic conditions and are able to complete physical, cognitive, and psychosocial assessments. Recruitment will emphasize diversity, including racial/ethnic minority groups and individuals from underserved communities, with study materials available in English and Spanish.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in adherence to Health Passport recommendations-Physical/Cardiovascular Health (HPAI-PC) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Adherence Index (HPAI) Physical/Cardiovascular health; study-specific index. 5-item Likert index (0-4 per item), domain total 0-20; higher = better adherence. Unit: points.
Change in adherence to Health Passport recommendations-Cognitive, Sleep, and Mental Health (HPAI-CSM) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Adherence Index (HPAI) for Cognitive, Sleep and Mental Health. 5-item Likert index (0-4 per item), domain total 0-20; higher = better adherence. Unit: points.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  The Montreal Cognitive Assessment (MoCA) is a 30-point scale used to assess global cognitive function, including memory, attention, language, and executive function. Higher scores indicate better cognitive performance.
Change in static balance (Four-Stage Balance Test) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Total seconds successfully held across 4 stances (0-40 s); higher = better. Unit: seconds.
Change in adherence to Health Passport recommendations-Diet and Oral Health (HPAI-DO) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Adherence Index (HPAI) Diet and Oral Health. 5-item Likert index (0-4 per item), domain total 0-20; higher = better adherence. Unit: points.
Change in adherence to Health Passport recommendations-Social Health (HPAI-SH) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Adherence Index (HPAI) for Social Health. 5-item Likert index (0-4 per item), domain total 0-20; higher = better adherence. Unit: points.
Change in walking endurance (200-Meter Fast Walk Test) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Seconds to complete 200 m at fastest safe pace; lower = better. Unit: seconds.
Change in gait speed (10-Meter Walk Test) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Comfortable-pace gait speed over 10 m; meters/second; higher = better. Unit: m/s.
Change in PROMIS-57 Sleep Disturbance | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 Sleep Disturbance T-score (mean 50, SD 10); higher = worse. Unit: T-score.
Change in PROMIS-57 Pain Interference | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 (Patient-Reported Outcomes Measurement Information System.) Pain Interference T-score (mean 50, SD 10); higher = worse. Unit: T-score.
Change in PROMIS-57 Fatigue | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 Fatigue T-score (mean 50, SD 10); higher = worse. Unit: T-score.
Change in PROMIS-57 Depression | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 Depression T-score (mean 50, SD 10); higher = worse. Unit: T-score.
Change in PROMIS-57 Anxiety | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 (Patient-Reported Outcomes Measurement Information System) Anxiety T-score (mean 50, SD 10); higher = worse. Unit: T-score.
Change in PROMIS-57 Satisfaction with Social Roles | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 Satisfaction with Social Roles T-score (mean 50, SD 10); higher = better. Unit: T-score.
Change in PROMIS-57 Physical Function | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  PROMIS-57 (Patient-Reported Outcomes Measurement Information System) Physical Function T-score (mean 50, SD 10); higher = better function. Unit: T-score.
Change in depressive symptoms (CES-D-20) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Center for Epidemiologic Studies Depression Scale-20 items (0-3 per item based on past-week frequency: 0=rarely/none, 1=some/a little, 2=occasionally/moderate, 3=most/all); total 0-60; higher = worse depressive symptoms. Unit: points.
Change in self-reported cognitive function (Neuro-QOL v2.0 Cognitive Function) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Neuro-QOL (Quality of Life in Neurological Disorders) Cognitive Function T-score (mean 50, SD 10); higher = better cognitive function. Unit: T-score.
Change in falls incidence (self-report) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Number of falls in the prior 12 months, self-reported. Unit: number of falls. Fewer falls indicates a better outcome.
Change in Central Nervous System (CNS) Vital Signs composite scores | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  CNS Vital Signs is a computerized neurocognitive test battery that evaluates domains such as memory, attention, executive function, and processing speed. Scores are standardized (mean = 100, SD = 15) and age-matched, with higher scores reflecting better function.
Change in systolic and diastolic blood pressure | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Resting systolic and diastolic blood pressure will be measured in millimeters of mercury (mmHg) using a standardized sphygmomanometer.
Change in body composition (bioimpedance) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Body composition will be measured using bioelectrical impedance analysis, reporting the percentage (%) body fat and kilograms (kg) lean tissue mass.
Change in MIND Diet Score | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  The MIND (Mediterranean-DASH Intervention for Neurodegenerative Delay) Diet Score measures adherence to dietary patterns associated with reduced risk of cognitive decline. Scores are based on frequency of consumption of 15 food groups. The total score ranges from 0 to 15, with higher scores indicating greater adherence to the MIND diet and better diet quality.
Change in Timed Up and Go (TUG) test scores | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  The Timed Up and Go test measures functional mobility. Participants are timed while standing up from a chair, walking 3 meters, turning, walking back, and sitting down. Lower times indicate better mobility.
Change in 6-Minute Walk Test distance | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  The 6-Minute Walk Test measures functional exercise capacity by recording the distance an individual can walk in 6 minutes on a flat surface. Greater distances, measured in meters (m), indicate better mobility and endurance.
Change in Body Mass Index (BMI) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  BMI (kg/m²); numeric measure; interpretation relative to clinical ranges. In most cases, "better" scores are indicated by closer proximity to normal BMI (18.5-24.5), with lower scores indicating an underweight BMI and higher scores indicating an overweight BMI. Unit: kg/m².
Change in oral-health-related quality of life (GOHAI) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Geriatric Oral Health Assessment Index (GOHAI); Score range is 12-60; higher = better oral-health-related quality of life. Unit: points.
Change in perceived stress (A-SDH) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Perceived Stress construct standardized score per A-SDH (All of Us Social Determinants of Health) scoring per U.S. Department of Health and Human Services; higher score = worse stress. Unit: standardized construct score.

OTHER OUTCOMES:
Change in food insecurity (A-SDH) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Proportion of participants screening positive for food insecurity (All of Us Social Determinants of Health, from the U.S. Department of Health and Human Services); lower proportion = better. Unit: percent of participants.
Change in transportation difficulty (A-SDH) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Proportion of participants endorsing transportation barriers, per the A-SDH (All of Us Social Determinants of Health, from the U.S. Department of Health and Human Services); lower proportion = better. Unit: percent of participants.
Overall adherence to Health Passport recommendations (HPAI total; exploratory) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Sum of the four Health Passport Adherence Index (HPAI) domain scores (0-80). If one domain is N/A, average available domains and multiply by 4. Higher = better adherence. Unit: points.
Change in Health Passport usability (HPUS; exploratory) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Usability Score (HPUS), 5-item Likert index (0-4 per item). Items: usefulness, clarity, ease of following, goal-setting support, sharing frequency (Likert). Total 0-20; higher = better usability. Unit: points.
Change in arterial stiffness (arteriography) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Arterial stiffness will be assessed by pulse wave velocity (PWV), measured in meters per second or via a comparable arteriography method. Higher values indicate greater stiffness.
Change in resting heart rate | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Resting heart rate (measured in beats per minute [bpm]) will be measured after 5 minutes of seated rest.
Change in Health Passport Usability Score (HPUS) | Baseline and 12 months (with annual re-testing up to 5 years, per protocol).
  Health Passport Usability Score (HPUS), a 5 item Likert index. Each item scored 0-4 (0=strongly disagree, 1=disagree, 2=neither agree nor disagree, 3=agree, 4=strongly agree). Total 0-20; higher scores indicate better usability. Unit: points.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Heyn, PhD, FGSA, FACRM, Principal Investigator — Office of Research, Marymount University
Locations (1):
- Center for Optimal Aging, Marymount University, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD used for the resulting publication(s) will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available immediately following the publication of study results. Results will be made available indefinitely via an appropriate public repository.

REFERENCES:
- [Background] Blank K, Gruman C, Robison JT. Case-finding for depression in elderly people: balancing ease of administration with validity in varied treatment settings. J Gerontol A Biol Sci Med Sci. 2004 Apr;59(4):378-84. doi: 10.1093/gerona/59.4.m378. PMID 15071082
- [Background] Ng TKS, Coughlan C, Heyn PC, Tagawa A, Carollo JJ, Kua EH, Mahendran R. Increased plasma brain-derived neurotrophic factor (BDNF) as a potential biomarker for and compensatory mechanism in mild cognitive impairment: a case-control study. Aging (Albany NY). 2021 Oct 15;13(19):22666-22689. doi: 10.18632/aging.203598. Epub 2021 Oct 15. PMID 34607976
- [Background] MacCarthy M, Heyn P, Tagawa A, Carollo J. Walking speed and patient-reported outcomes in young adults with cerebral palsy. Dev Med Child Neurol. 2022 Oct;64(10):1281-1288. doi: 10.1111/dmcn.15225. Epub 2022 Apr 2. PMID 35366333
- [Background] Hegarty, M., Montello, D. R., Richardson, A. E., Ishikawa, T., & Lovelace, K. (2006). Spatial abilities at different scales: Individual differences in aptitude-test performance and spatial-layout learning. Intelligence, 34(2), 151-176. https://doi.org/10.1016/j.intell.2005.09.005
- [Background] Olabarrieta-Landa L, Rivera D, Galarza-Del-Angel J, Garza MT, Saracho CP, Rodriguez W, Chavez-Oliveros M, Rabago B, Leibach G, Schebela S, Martinez C, Luna M, Longoni M, Ocampo-Barba N, Rodriguez G, Aliaga A, Esenarro L, Garcia de la Cadena C, Perrin BP, Arango-Lasprilla JC. Verbal fluency tests: Normative data for the Latin American Spanish speaking adult population. NeuroRehabilitation. 2015;37(4):515-61. doi: 10.3233/NRE-151279. PMID 26639930
- [Background] Hurtado-Pomares M, Juarez-Leal I, Company-Devesa V, Sanchez-Perez A, Peral-Gomez P, Espinosa-Sempere C, Valera-Gran D, Navarrete-Munoz EM. Psychometric properties of the Spanish version of the Frontal Assessment Battery (FAB-E) and normative values in a representative adult population sample. Neurologia (Engl Ed). 2024 Oct;39(8):694-700. doi: 10.1016/j.nrleng.2022.09.004. Epub 2022 Oct 7. PMID 36216225
- [Background] Arango-Lasprilla JC, Rivera D, Aguayo A, Rodriguez W, Garza MT, Saracho CP, Rodriguez-Agudelo Y, Aliaga A, Weiler G, Luna M, Longoni M, Ocampo-Barba N, Galarza-Del-Angel J, Panyavin I, Guerra A, Esenarro L, Garcia de la Cadena P, Martinez C, Perrin PB. Trail Making Test: Normative data for the Latin American Spanish speaking adult population. NeuroRehabilitation. 2015;37(4):639-61. doi: 10.3233/NRE-151284. PMID 26639932
- [Background] Gollan TH, Garcia DL, Stasenko A, Murillo M, Kim C, Galasko D, Salmon DP. The MINT Sprint 2.0: A picture naming test for detection of naming impairments in Alzheimer's disease and in preclinical AD. Alzheimers Dement. 2024 Jan;20(1):112-123. doi: 10.1002/alz.13381. Epub 2023 Jul 19. PMID 37464962
- [Background] He Z, Dieciuc M, Carr D, Chakraborty S, Singh A, Fowe IE, Zhang S, Lustria MLA, Terracciano A, Charness N, Boot WR. New Opportunities for the Early Detection and Treatment of Cognitive Decline: Adherence Challenges and the Promise of Smart and Person-Centered Technologies. BMC Digit Health. 2023;1:7. doi: 10.1186/s44247-023-00008-1. Epub 2023 Feb 14. PMID 40093660
- [Background] Olivari BS, Baumgart M, Lock SL, Whiting CG, Taylor CA, Iskander J, Thorpe P, McGuire LC. CDC Grand Rounds: Promoting Well-Being and Independence in Older Adults. MMWR Morb Mortal Wkly Rep. 2018 Sep 21;67(37):1036-1039. doi: 10.15585/mmwr.mm6737a4. PMID 30235185
- [Background] Visscher TL, Seidell JC, Molarius A, van der Kuip D, Hofman A, Witteman JC. A comparison of body mass index, waist-hip ratio and waist circumference as predictors of all-cause mortality among the elderly: the Rotterdam study. Int J Obes Relat Metab Disord. 2001 Nov;25(11):1730-5. doi: 10.1038/sj.ijo.0801787. PMID 11753597
- [Background] Ma W, Zhu H, Yu X, Zhai X, Li S, Huang N, Liu K, Shirai K, Sheerah HA, Cao J. Association between android fat mass, gynoid fat mass and cardiovascular and all-cause mortality in adults: NHANES 2003-2007. Front Cardiovasc Med. 2023 May 18;10:1055223. doi: 10.3389/fcvm.2023.1055223. eCollection 2023. PMID 37273879
- [Background] Abellan van Kan G, Rolland Y, Andrieu S, Bauer J, Beauchet O, Bonnefoy M, Cesari M, Donini LM, Gillette Guyonnet S, Inzitari M, Nourhashemi F, Onder G, Ritz P, Salva A, Visser M, Vellas B. Gait speed at usual pace as a predictor of adverse outcomes in community-dwelling older people an International Academy on Nutrition and Aging (IANA) Task Force. J Nutr Health Aging. 2009 Dec;13(10):881-9. doi: 10.1007/s12603-009-0246-z. PMID 19924348
- [Background] Bohannon RW. Reference values for the timed up and go test: a descriptive meta-analysis. J Geriatr Phys Ther. 2006;29(2):64-8. doi: 10.1519/00139143-200608000-00004. PMID 16914068
- [Background] Rossiter-Fornoff JE, Wolf SL, Wolfson LI, Buchner DM. A cross-sectional validation study of the FICSIT common data base static balance measures. Frailty and Injuries: Cooperative Studies of Intervention Techniques. J Gerontol A Biol Sci Med Sci. 1995 Nov;50(6):M291-7. doi: 10.1093/gerona/50a.6.m291. PMID 7583799
- [Background] Bohannon RW. Grip Strength: An Indispensable Biomarker For Older Adults. Clin Interv Aging. 2019 Oct 1;14:1681-1691. doi: 10.2147/CIA.S194543. eCollection 2019. PMID 31631989
- [Background] Gates DH, Walters LS, Cowley J, Wilken JM, Resnik L. Range of Motion Requirements for Upper-Limb Activities of Daily Living. Am J Occup Ther. 2016 Jan-Feb;70(1):7001350010p1-7001350010p10. doi: 10.5014/ajot.2016.015487. PMID 26709433
- [Background] Bhattacharya, P. (n.d.). Assessment of inter-rater variability of the Senior Fitness Test in the geriatric population: A community based study. ResearchGate. Retrieved October 28, 2024, from https://www.researchgate.net/publication/311446863_Assessment_of_inter-rater_variability_of_the_Senior_Fitness_Test_in_the_geriatric_population_A_community_based_study
- [Background] Straight CR, Dorfman LR, Cottell KE, Krol JM, Lofgren IE, Delmonico MJ. Effects of resistance training and dietary changes on physical function and body composition in overweight and obese older adults. J Phys Act Health. 2012 Aug;9(6):875-83. doi: 10.1123/jpah.9.6.875. Epub 2011 Aug 2. PMID 21952180
- [Background] Lynall RC, Zukowski LA, Plummer P, Mihalik JP. Reliability and validity of the protokinetics movement analysis software in measuring center of pressure during walking. Gait Posture. 2017 Feb;52:308-311. doi: 10.1016/j.gaitpost.2016.12.023. Epub 2016 Dec 21. PMID 28033577
- [Background] Wang KL, Cheng HM, Sung SH, Chuang SY, Li CH, Spurgeon HA, Ting CT, Najjar SS, Lakatta EG, Yin FC, Chou P, Chen CH. Wave reflection and arterial stiffness in the prediction of 15-year all-cause and cardiovascular mortalities: a community-based study. Hypertension. 2010 Mar;55(3):799-805. doi: 10.1161/HYPERTENSIONAHA.109.139964. Epub 2010 Jan 11. PMID 20065155
- [Background] Roman MJ, Devereux RB, Kizer JR, Lee ET, Galloway JM, Ali T, Umans JG, Howard BV. Central pressure more strongly relates to vascular disease and outcome than does brachial pressure: the Strong Heart Study. Hypertension. 2007 Jul;50(1):197-203. doi: 10.1161/HYPERTENSIONAHA.107.089078. Epub 2007 May 7. PMID 17485598
- [Background] McEniery CM, Cockcroft JR, Roman MJ, Franklin SS, Wilkinson IB. Central blood pressure: current evidence and clinical importance. Eur Heart J. 2014 Jul;35(26):1719-25. doi: 10.1093/eurheartj/eht565. Epub 2014 Jan 23. PMID 24459197
- [Background] Vlachopoulos C, Aznaouridis K, O'Rourke MF, Safar ME, Baou K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with central haemodynamics: a systematic review and meta-analysis. Eur Heart J. 2010 Aug;31(15):1865-71. doi: 10.1093/eurheartj/ehq024. Epub 2010 Mar 2. PMID 20197424
- [Background] Lakatta EG. Arterial and cardiac aging: major shareholders in cardiovascular disease enterprises: Part III: cellular and molecular clues to heart and arterial aging. Circulation. 2003 Jan 28;107(3):490-7. doi: 10.1161/01.cir.0000048894.99865.02. No abstract available. PMID 12551876
- [Background] Munir S, Jiang B, Guilcher A, Brett S, Redwood S, Marber M, Chowienczyk P. Exercise reduces arterial pressure augmentation through vasodilation of muscular arteries in humans. Am J Physiol Heart Circ Physiol. 2008 Apr;294(4):H1645-50. doi: 10.1152/ajpheart.01171.2007. Epub 2008 Feb 22. PMID 18296568
- [Background] Nichols WW. Clinical measurement of arterial stiffness obtained from noninvasive pressure waveforms. Am J Hypertens. 2005 Jan;18(1 Pt 2):3S-10S. doi: 10.1016/j.amjhyper.2004.10.009. PMID 15683725
- [Background] Vlachopoulos C, Xaplanteris P, Aboyans V, Brodmann M, Cifkova R, Cosentino F, De Carlo M, Gallino A, Landmesser U, Laurent S, Lekakis J, Mikhailidis DP, Naka KK, Protogerou AD, Rizzoni D, Schmidt-Trucksass A, Van Bortel L, Weber T, Yamashina A, Zimlichman R, Boutouyrie P, Cockcroft J, O'Rourke M, Park JB, Schillaci G, Sillesen H, Townsend RR. The role of vascular biomarkers for primary and secondary prevention. A position paper from the European Society of Cardiology Working Group on peripheral circulation: Endorsed by the Association for Research into Arterial Structure and Physiology (ARTERY) Society. Atherosclerosis. 2015 Aug;241(2):507-32. doi: 10.1016/j.atherosclerosis.2015.05.007. Epub 2015 May 16. PMID 26117398
- [Background] Laurent S, Boutouyrie P, Asmar R, Gautier I, Laloux B, Guize L, Ducimetiere P, Benetos A. Aortic stiffness is an independent predictor of all-cause and cardiovascular mortality in hypertensive patients. Hypertension. 2001 May;37(5):1236-41. doi: 10.1161/01.hyp.37.5.1236. PMID 11358934
- [Background] O'Rourke MF, Staessen JA, Vlachopoulos C, Duprez D, Plante GE. Clinical applications of arterial stiffness; definitions and reference values. Am J Hypertens. 2002 May;15(5):426-44. doi: 10.1016/s0895-7061(01)02319-6. PMID 12022246
- [Background] Boutouyrie P, Tropeano AI, Asmar R, Gautier I, Benetos A, Lacolley P, Laurent S. Aortic stiffness is an independent predictor of primary coronary events in hypertensive patients: a longitudinal study. Hypertension. 2002 Jan;39(1):10-5. doi: 10.1161/hy0102.099031. PMID 11799071
- [Background] Zota IM, Statescu C, Sascau RA, Roca M, Anghel L, Mitu O, Ghiciuc CM, Boisteanu D, Anghel R, Cozma SR, Dima-Cozma LC, Mitu F. Arterial Stiffness Assessment Using the Arteriograph in Patients with Moderate-Severe OSA and Metabolic Syndrome-A Pilot Study. J Clin Med. 2021 Sep 18;10(18):4238. doi: 10.3390/jcm10184238. PMID 34575349
- [Background] Beckman JA, Higgins CO, Gerhard-Herman M. Automated oscillometric determination of the ankle-brachial index provides accuracy necessary for office practice. Hypertension. 2006 Jan;47(1):35-8. doi: 10.1161/01.HYP.0000196686.85286.9c. Epub 2005 Dec 12. PMID 16344373
- [Background] O'Brien E, Petrie J, Littler W, de Swiet M, Padfield PL, O'Malley K, Jamieson M, Altman D, Bland M, Atkins N. The British Hypertension Society protocol for the evaluation of automated and semi-automated blood pressure measuring devices with special reference to ambulatory systems. J Hypertens. 1990 Jul;8(7):607-19. doi: 10.1097/00004872-199007000-00004. PMID 2168451
- [Background] Fulbrook P. Core body temperature measurement: a comparison of axilla, tympanic membrane and pulmonary artery blood temperature. Intensive Crit Care Nurs. 1997 Oct;13(5):266-72. doi: 10.1016/s0964-3397(97)80425-9. PMID 9538713
- [Background] Borg, G. (1998). Borg's perceived exertion and pain scales (pp. viii, 104). Human Kinetics.
- [Background] Aguirre-Bustamante J, Baron-Lopez FJ, Carmona-Gonzalez FJ, Perez-Farinos N, Warnberg J. Validation of a modified version of the Spanish Geriatric Oral Health Assessment Index (GOHAI-SP) for adults and elder people. BMC Oral Health. 2020 Feb 19;20(1):61. doi: 10.1186/s12903-020-1047-3. PMID 32075623
- [Background] Wright FAC, Law G, Chu SK, Cullen JS, Le Couteur DG. Residential age care and domiciliary oral health services: Reach-OHT-The development of a metropolitan oral health programme in Sydney, Australia. Gerodontology. 2017 Dec;34(4):420-426. doi: 10.1111/ger.12282. Epub 2017 Jul 19. PMID 28722250
- [Background] Aguilar-Navarro SG, Mimenza-Alvarado AJ, Palacios-Garcia AA, Samudio-Cruz A, Gutierrez-Gutierrez LA, Avila-Funes JA. Validity and Reliability of the Spanish Version of the Montreal Cognitive Assessment (MoCA) for the Detection of Cognitive Impairment in Mexico. Rev Colomb Psiquiatr (Engl Ed). 2018 Oct-Dec;47(4):237-243. doi: 10.1016/j.rcp.2017.05.003. Epub 2017 Jul 29. English, Spanish. PMID 30286846
- [Background] Apiquian R, Diaz R, Victoria G, Ulloa RE. The Category Fluency Test components and their association with cognition and symptoms in adolescents with schizophrenia. Schizophr Res Cogn. 2023 Nov 10;35:100296. doi: 10.1016/j.scog.2023.100296. eCollection 2024 Mar. PMID 38025823
- [Background] Hassel AJ, Rolko C, Koke U, Leisen J, Rammelsberg P. A German version of the GOHAI. Community Dent Oral Epidemiol. 2008 Feb;36(1):34-42. doi: 10.1111/j.1600-0528.2007.00351.x. PMID 18205638
- [Background] Rubenstein LZ, Vivrette R, Harker JO, Stevens JA, Kramer BJ. Validating an evidence-based, self-rated fall risk questionnaire (FRQ) for older adults. J Safety Res. 2011 Dec;42(6):493-9. doi: 10.1016/j.jsr.2011.08.006. Epub 2011 Nov 17. PMID 22152267
- [Background] Anton SD, Woods AJ, Ashizawa T, Barb D, Buford TW, Carter CS, Clark DJ, Cohen RA, Corbett DB, Cruz-Almeida Y, Dotson V, Ebner N, Efron PA, Fillingim RB, Foster TC, Gundermann DM, Joseph AM, Karabetian C, Leeuwenburgh C, Manini TM, Marsiske M, Mankowski RT, Mutchie HL, Perri MG, Ranka S, Rashidi P, Sandesara B, Scarpace PJ, Sibille KT, Solberg LM, Someya S, Uphold C, Wohlgemuth S, Wu SS, Pahor M. Successful aging: Advancing the science of physical independence in older adults. Ageing Res Rev. 2015 Nov;24(Pt B):304-27. doi: 10.1016/j.arr.2015.09.005. Epub 2015 Oct 14. PMID 26462882
- [Background] Mahmood SS, Levy D, Vasan RS, Wang TJ. The Framingham Heart Study and the epidemiology of cardiovascular disease: a historical perspective. Lancet. 2014 Mar 15;383(9921):999-1008. doi: 10.1016/S0140-6736(13)61752-3. Epub 2013 Sep 29. PMID 24084292
- [Background] Kivipelto M, Mangialasche F, Snyder HM, Allegri R, Andrieu S, Arai H, Baker L, Belleville S, Brodaty H, Brucki SM, Calandri I, Caramelli P, Chen C, Chertkow H, Chew E, Choi SH, Chowdhary N, Crivelli L, Torre R, Du Y, Dua T, Espeland M, Feldman HH, Hartmanis M, Hartmann T, Heffernan M, Henry CJ, Hong CH, Hakansson K, Iwatsubo T, Jeong JH, Jimenez-Maggiora G, Koo EH, Launer LJ, Lehtisalo J, Lopera F, Martinez-Lage P, Martins R, Middleton L, Molinuevo JL, Montero-Odasso M, Moon SY, Morales-Perez K, Nitrini R, Nygaard HB, Park YK, Peltonen M, Qiu C, Quiroz YT, Raman R, Rao N, Ravindranath V, Rosenberg A, Sakurai T, Salinas RM, Scheltens P, Sevlever G, Soininen H, Sosa AL, Suemoto CK, Tainta-Cuezva M, Velilla L, Wang Y, Whitmer R, Xu X, Bain LJ, Solomon A, Ngandu T, Carrillo MC. World-Wide FINGERS Network: A global approach to risk reduction and prevention of dementia. Alzheimers Dement. 2020 Jul;16(7):1078-1094. doi: 10.1002/alz.12123. Epub 2020 Jul 5. PMID 32627328
- [Background] Jack CR Jr, Albert MS, Knopman DS, McKhann GM, Sperling RA, Carrillo MC, Thies B, Phelps CH. Introduction to the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):257-62. doi: 10.1016/j.jalz.2011.03.004. Epub 2011 Apr 21. PMID 21514247
- [Background] Stanziano DC, Whitehurst M, Graham P, Roos BA. A review of selected longitudinal studies on aging: past findings and future directions. J Am Geriatr Soc. 2010 Oct;58 Suppl 2(Suppl 2):S292-7. doi: 10.1111/j.1532-5415.2010.02936.x. PMID 21029056
- [Background] Caruana EJ, Roman M, Hernandez-Sanchez J, Solli P. Longitudinal studies. J Thorac Dis. 2015 Nov;7(11):E537-40. doi: 10.3978/j.issn.2072-1439.2015.10.63. No abstract available. PMID 26716051
- [Background] Tangney CC, Li H, Wang Y, Barnes L, Schneider JA, Bennett DA, Morris MC. Relation of DASH- and Mediterranean-like dietary patterns to cognitive decline in older persons. Neurology. 2014 Oct 14;83(16):1410-6. doi: 10.1212/WNL.0000000000000884. Epub 2014 Sep 17. PMID 25230996
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Kramarow EA. Dental Care Among Adults Aged 65 and Over, 2017. NCHS Data Brief. 2019 May;(337):1-8. PMID 31163014
- [Background] Wilentz JB, Kleinman DV, Alfano MC. Meeting commentary: Santa Fe Group Salon Expanding Oral Healthcare for America's Seniors, September 28-30, 2016. J Am Dent Assoc. 2017 Apr;148(4):272-274. doi: 10.1016/j.adaj.2017.01.028. PMID 28359455
- [Background] Cristina NM, Lucia D. Nutrition and Healthy Aging: Prevention and Treatment of Gastrointestinal Diseases. Nutrients. 2021 Nov 30;13(12):4337. doi: 10.3390/nu13124337. PMID 34959889
- [Background] Noble JM, Borrell LN, Papapanou PN, Elkind MS, Scarmeas N, Wright CB. Periodontitis is associated with cognitive impairment among older adults: analysis of NHANES-III. J Neurol Neurosurg Psychiatry. 2009 Nov;80(11):1206-11. doi: 10.1136/jnnp.2009.174029. Epub 2009 May 5. PMID 19419981
- [Background] Moriya S, Tei K, Murata A, Yamazaki Y, Hata H, Muramatsu M, Kitagawa Y, Inoue N, Miura H. Associations between self-assessed masticatory ability and higher brain function among the elderly. J Oral Rehabil. 2011 Oct;38(10):746-53. doi: 10.1111/j.1365-2842.2011.02214.x. Epub 2011 Mar 23. PMID 21428989
- [Background] Lin CS. Revisiting the link between cognitive decline and masticatory dysfunction. BMC Geriatr. 2018 Jan 5;18(1):5. doi: 10.1186/s12877-017-0693-z. PMID 29304748
- [Background] Dintica CS, Marseglia A, Wardh I, Stjernfeldt Elgestad P, Rizzuto D, Shang Y, Xu W, Pedersen NL. The relation of poor mastication with cognition and dementia risk: a population-based longitudinal study. Aging (Albany NY). 2020 Apr 30;12(9):8536-8548. doi: 10.18632/aging.103156. Epub 2020 Apr 30. PMID 32353829
- [Background] Raphael C. Oral Health and Aging. Am J Public Health. 2017 May;107(S1):S44-S45. doi: 10.2105/AJPH.2017.303835. No abstract available. PMID 28661797
- [Background] Ahlskog JE, Geda YE, Graff-Radford NR, Petersen RC. Physical exercise as a preventive or disease-modifying treatment of dementia and brain aging. Mayo Clin Proc. 2011 Sep;86(9):876-84. doi: 10.4065/mcp.2011.0252. PMID 21878600
- [Background] Feito, Y. (n.d.). ACSM's Guidelines for Exercise Testing and Prescription. Retrieved October 28, 2024, from https://www.wolterskluwer.com/en/know/acsm/guidelines-for-exercise-testing-and-prescription
- [Background] Cicalese SM, da Silva JF, Priviero F, Webb RC, Eguchi S, Tostes RC. Vascular Stress Signaling in Hypertension. Circ Res. 2021 Apr 2;128(7):969-992. doi: 10.1161/CIRCRESAHA.121.318053. Epub 2021 Apr 1. PMID 33793333
- [Background] Anisimova AS, Alexandrov AI, Makarova NE, Gladyshev VN, Dmitriev SE. Protein synthesis and quality control in aging. Aging (Albany NY). 2018 Dec 18;10(12):4269-4288. doi: 10.18632/aging.101721. PMID 30562164
- [Background] Yi Y, Baek JY, Lee E, Jung HW, Jang IY. A Comparative Study of High-Frequency Bioelectrical Impedance Analysis and Dual-Energy X-ray Absorptiometry for Estimating Body Composition. Life (Basel). 2022 Jul 4;12(7):994. doi: 10.3390/life12070994. PMID 35888083
- [Background] Timmerman KL, Dhanani S, Glynn EL, Fry CS, Drummond MJ, Jennings K, Rasmussen BB, Volpi E. A moderate acute increase in physical activity enhances nutritive flow and the muscle protein anabolic response to mixed nutrient intake in older adults. Am J Clin Nutr. 2012 Jun;95(6):1403-12. doi: 10.3945/ajcn.111.020800. Epub 2012 May 9. PMID 22572647
- [Background] Ruiz JG, Dent E, Morley JE, Merchant RA, Beilby J, Beard J, Tripathy C, Sorin M, Andrieu S, Aprahamian I, Arai H, Aubertin-Leheudre M, Bauer JM, Cesari M, Chen LK, Cruz-Jentoft AJ, De Souto Barreto P, Dong B, Ferrucci L, Fielding R, Flicker L, Lundy J, Reginster JY, Rodriguez-Manas L, Rolland Y, Sanford AM, Sinclair AJ, Vina J, Waters DL, Won Won C, Woo J, Vellas B. Screening for and Managing the Person with Frailty in Primary Care: ICFSR Consensus Guidelines. J Nutr Health Aging. 2020;24(9):920-927. doi: 10.1007/s12603-020-1492-3. No abstract available. PMID 33155616
- [Background] Dent E, Martin FC, Bergman H, Woo J, Romero-Ortuno R, Walston JD. Management of frailty: opportunities, challenges, and future directions. Lancet. 2019 Oct 12;394(10206):1376-1386. doi: 10.1016/S0140-6736(19)31785-4. PMID 31609229
- [Background] Xue QL. The frailty syndrome: definition and natural history. Clin Geriatr Med. 2011 Feb;27(1):1-15. doi: 10.1016/j.cger.2010.08.009. PMID 21093718
- [Background] Gordon SJ, Baker N, Kidd M, Maeder A, Grimmer KA. Pre-frailty factors in community-dwelling 40-75 year olds: opportunities for successful ageing. BMC Geriatr. 2020 Mar 6;20(1):96. doi: 10.1186/s12877-020-1490-7. PMID 32143634
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Walston JD. Sarcopenia in older adults. Curr Opin Rheumatol. 2012 Nov;24(6):623-7. doi: 10.1097/BOR.0b013e328358d59b. PMID 22955023
- [Background] Fong JH. Disability incidence and functional decline among older adults with major chronic diseases. BMC Geriatr. 2019 Nov 21;19(1):323. doi: 10.1186/s12877-019-1348-z. PMID 31752701
- [Background] Ratnayake M; LPCMH; ATR; NCC;1; Lukas S, Brathwaite S, Neave J, Henry H; BS-c;5. Aging in Place:: Are We Prepared? Dela J Public Health. 2022 Aug 31;8(3):28-31. doi: 10.32481/djph.2022.08.007. eCollection 2022 Aug. PMID 36177171
- [Background] Office of Policy Development and Research. (n.d.). Measuring the Costs and Savings of Aging in Place HUD USER. Retrieved October 28, 2024, from
- [Background] Seider TR, Fieo RA, O'Shea A, Porges EC, Woods AJ, Cohen RA. Cognitively Engaging Activity Is Associated with Greater Cortical and Subcortical Volumes. Front Aging Neurosci. 2016 May 2;8:94. doi: 10.3389/fnagi.2016.00094. eCollection 2016. PMID 27199740
- [Background] Morris MC. Diet and Alzheimer's disease: what the evidence shows. MedGenMed. 2004 Jan 15;6(1):48. PMID 15208559
- [Background] Zhang XX, Tian Y, Wang ZT, Ma YH, Tan L, Yu JT. The Epidemiology of Alzheimer's Disease Modifiable Risk Factors and Prevention. J Prev Alzheimers Dis. 2021;8(3):313-321. doi: 10.14283/jpad.2021.15. PMID 34101789
- [Background] Committee on the Public Health Dimensions of Cognitive Aging; Board on Health Sciences Policy; Institute of Medicine; Blazer DG, Yaffe K, Liverman CT, editors. Cognitive Aging: Progress in Understanding and Opportunities for Action. Washington (DC): National Academies Press (US); 2015 Jul 21. Available from http://www.ncbi.nlm.nih.gov/books/NBK285319/ PMID 25879131
- [Background] Lopez-Ortiz S, Valenzuela PL, Seisdedos MM, Morales JS, Vega T, Castillo-Garcia A, Nistico R, Mercuri NB, Lista S, Lucia A, Santos-Lozano A. Exercise interventions in Alzheimer's disease: A systematic review and meta-analysis of randomized controlled trials. Ageing Res Rev. 2021 Dec;72:101479. doi: 10.1016/j.arr.2021.101479. Epub 2021 Sep 30. PMID 34601135
- [Background] Heyn PC, Johnson KE, Kramer AF. Endurance and strength training outcomes on cognitively impaired and cognitively intact older adults: a meta-analysis. J Nutr Health Aging. 2008 Jun-Jul;12(6):401-9. doi: 10.1007/BF02982674. PMID 18548179
- [Background] Etnier, J. L., Salazar, W., Landers, D. M., Petruzzello, S. J., Han, M., & Nowell, P. (1997). The influence of physical fitness and exercise upon cognitive functioning: A meta-analysis. In Database of Abstracts of Reviews of Effects (DARE): Quality-assessed Reviews Internet. Centre for Reviews and Dissemination (UK). https://www.ncbi.nlm.nih.gov/books/NBK67031
- [Background] Livingston G, Huntley J, Liu KY, Costafreda SG, Selbaek G, Alladi S, Ames D, Banerjee S, Burns A, Brayne C, Fox NC, Ferri CP, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Nakasujja N, Rockwood K, Samus Q, Shirai K, Singh-Manoux A, Schneider LS, Walsh S, Yao Y, Sommerlad A, Mukadam N. Dementia prevention, intervention, and care: 2024 report of the Lancet standing Commission. Lancet. 2024 Aug 10;404(10452):572-628. doi: 10.1016/S0140-6736(24)01296-0. Epub 2024 Jul 31. No abstract available. PMID 39096926
- [Background] Murman DL. The Impact of Age on Cognition. Semin Hear. 2015 Aug;36(3):111-21. doi: 10.1055/s-0035-1555115. PMID 27516712
- [Background] CDC. (2024, May 24). Preventing Chronic Diseases: What You Can Do Now. Chronic Disease. https://www.cdc.gov/chronic-disease/prevention/index.html
- [Background] Israel BA, Coombe CM, Cheezum RR, Schulz AJ, McGranaghan RJ, Lichtenstein R, Reyes AG, Clement J, Burris A. Community-based participatory research: a capacity-building approach for policy advocacy aimed at eliminating health disparities. Am J Public Health. 2010 Nov;100(11):2094-102. doi: 10.2105/AJPH.2009.170506. Epub 2010 Sep 23. PMID 20864728
- [Background] CDC. (2024, September 30). National Healthy Brain Initiative State and Local Road Map. Alzheimer's Disease Program. https://www.cdc.gov/aging-programs/php/nhbi/roadmap.html
- [Background] Administration for Community Living. (n.d.). 2021 Profile of Older Americans.
- [Background] National Academies of Sciences, Engineering, and Medicine; Division of Behavioral and Social Sciences and Education; Health and Medicine Division; Board on Behavioral, Cognitive, and Sensory Sciences; Board on Health Sciences Policy; Committee on the Health and Medical Dimensions of Social Isolation and Loneliness in Older Adults. Social Isolation and Loneliness in Older Adults: Opportunities for the Health Care System. Washington (DC): National Academies Press (US); 2020 Feb 27. Available from http://www.ncbi.nlm.nih.gov/books/NBK557974/ PMID 32510896
- [Background] Bailey ZD, Krieger N, Agenor M, Graves J, Linos N, Bassett MT. Structural racism and health inequities in the USA: evidence and interventions. Lancet. 2017 Apr 8;389(10077):1453-1463. doi: 10.1016/S0140-6736(17)30569-X. PMID 28402827
- [Background] National Institute on Aging. (n.d.). Goal B: Better understand the effects of personal, interpersonal, and societal factors on aging, including the mechanisms through which these factors exert their effects. National Institute on Aging. Retrieved October 28, 2024, from https://www.nia.nih.gov/about/aging-strategic-directions-research/goal-behavioral-psychological-factors
- [Background] Heyn PC, Baumgardner CA, McLachlan L, Bodine C. Mixed-reality exercise effects on participation of individuals with spinal cord injuries and developmental disabilities: a pilot study. Top Spinal Cord Inj Rehabil. 2014 Fall;20(4):338-45. doi: 10.1310/sci2004-338. PMID 25477747
- [Background] Heyn P, Abreu BC, Ottenbacher KJ. The effects of exercise training on elderly persons with cognitive impairment and dementia: a meta-analysis. Arch Phys Med Rehabil. 2004 Oct;85(10):1694-704. doi: 10.1016/j.apmr.2004.03.019. PMID 15468033
- [Background] Heyn P. The effect of a multisensory exercise program on engagement, behavior, and selected physiological indexes in persons with dementia. Am J Alzheimers Dis Other Demen. 2003 Jul-Aug;18(4):247-51. doi: 10.1177/153331750301800409. PMID 12955790
- [Background] Ng TKS, Tagawa A, Ho RC, Larbi A, Kua EH, Mahendran R, Carollo JJ, Heyn PC. Commonalities in biomarkers and phenotypes between mild cognitive impairment and cerebral palsy: a pilot exploratory study. Aging (Albany NY). 2021 Jan 26;13(2):1773-1816. doi: 10.18632/aging.202563. Epub 2021 Jan 26. PMID 33497355
- [Background] Caselli RJ, Langlais BT, Dueck AC, Chen Y, Su Y, Locke DEC, Woodruff BK, Reiman EM. Neuropsychological decline up to 20 years before incident mild cognitive impairment. Alzheimers Dement. 2020 Mar;16(3):512-523. doi: 10.1016/j.jalz.2019.09.085. Epub 2020 Jan 6. PMID 31787561
- [Background] Glasgow RE, Vinson C, Chambers D, Khoury MJ, Kaplan RM, Hunter C. National Institutes of Health approaches to dissemination and implementation science: current and future directions. Am J Public Health. 2012 Jul;102(7):1274-81. doi: 10.2105/AJPH.2012.300755. Epub 2012 May 17. PMID 22594758
- [Background] Towfighi A, Orechwa AZ, Aragon TJ, Atkins M, Brown AF, Brown J, Carrasquillo O, Carson S, Fleisher P, Gustafson E, Herman DK, Inkelas M, Liu W, Meeker D, Mehta T, Miller DC, Paul-Brutus R, Potter MB, Ritner SS, Rodriguez B, Rusch D, Skinner A, Yee HF Jr. Bridging the gap between research, policy, and practice: Lessons learned from academic-public partnerships in the CTSA network. J Clin Transl Sci. 2020 Mar 10;4(3):201-208. doi: 10.1017/cts.2020.23. PMID 32695489
- [Background] Watson C. Many researchers say they'll share data - but don't. Nature. 2022 Jun;606(7916):853. doi: 10.1038/d41586-022-01692-1. No abstract available. PMID 35725829
- [Background] McKibbin KJ, Malin BA, Clayton EW. Protecting research data of publicly revealing participants. J Law Biosci. 2021 Sep 6;8(2):lsab028. doi: 10.1093/jlb/lsab028. eCollection 2021 Jul-Dec. PMID 34512997
- [Background] McElfish PA, Long CR, James LP, Scott AJ, Flood-Grady E, Kimminau KS, Rhyne RL, Burge MR, Purvis RS. Characterizing health researcher barriers to sharing results with study participants. J Clin Transl Sci. 2019 Oct 4;3(6):295-301. doi: 10.1017/cts.2019.409. eCollection 2019 Dec. PMID 31827902
- [Background] Long CR, Purvis RS, Flood-Grady E, Kimminau KS, Rhyne RL, Burge MR, Stewart MK, Jenkins AJ, James LP, McElfish PA. Health researchers' experiences, perceptions and barriers related to sharing study results with participants. Health Res Policy Syst. 2019 Mar 4;17(1):25. doi: 10.1186/s12961-019-0422-5. PMID 30832733
- [Background] Cherbuin N, Iijima K, Kalula S, Malhotra R, Rasmussen LJ, Chan A, Lafortune L, Harper S, Zheng X, Lindeman D, Walsh E, Hussain R, Burns R, Kristiansen M, Sugawara I, Son B, Tanaka T, Buckner S, Hoffman J, Combrinck M. Societal Need for Interdisciplinary Ageing Research: An International Alliance of Research Universities "Ageing, Longevity and Health" Stream (IARU-ALH) Position Statement. Biomed Hub. 2021 Feb 25;6(1):42-47. doi: 10.1159/000513513. eCollection 2021 Jan-Apr. PMID 33791316
- [Background] Stange KC. The problem of fragmentation and the need for integrative solutions. Ann Fam Med. 2009 Mar-Apr;7(2):100-3. doi: 10.1370/afm.971. No abstract available. PMID 19273863
- [Background] Kenneth Brummel-Smith, M. D. (2008). Optimal Aging, Part I: Demographics and Definitions. Annals of Long-Term Care, 15(11). https://www.hmpgloballearningnetwork.com/site/altc/article/7994
- [Background] Gurwitz JH. The Paradoxical Decline of Geriatric Medicine as a Profession. JAMA. 2023 Aug 22;330(8):693-694. doi: 10.1001/jama.2023.11110. PMID 37540519
- [Background] Chatterji S, Byles J, Cutler D, Seeman T, Verdes E. Health, functioning, and disability in older adults--present status and future implications. Lancet. 2015 Feb 7;385(9967):563-75. doi: 10.1016/S0140-6736(14)61462-8. Epub 2014 Nov 6. PMID 25468158
- [Background] World Health Organization. (n.d.). Life expectancy at birth (years). Retrieved October 28, 2024, from https://www.who.int/data/gho/data/indicators/indicator-details/GHO/life-expectancy-at-birth-(years)
- [Background] Peterson, T. (n.d.). Healthspan is more important than lifespan, so why don't more people know about it? Institute for Public Health Washington University in St. Louis. Retrieved October 28, 2024, from https://publichealth.wustl.edu/heatlhspan-is-more-important-than-lifespan-so-why-dont-more-people-know-about-it/
- [Background] Olshansky SJ. From Lifespan to Healthspan. JAMA. 2018 Oct 2;320(13):1323-1324. doi: 10.1001/jama.2018.12621. No abstract available. PMID 30242384
- [Background] White MC, Holman DM, Goodman RA, Richardson LC. Cancer Risk Among Older Adults: Time for Cancer Prevention to Go Silver. Gerontologist. 2019 Jun;59(Suppl 1):S1-S6. doi: 10.1093/geront/gnz038. Epub 2019 May 17. PMID 31511747
- [Background] Balasubramanian P, Kiss T, Tarantini S, Nyul-Toth A, Ahire C, Yabluchanskiy A, Csipo T, Lipecz A, Tabak A, Institoris A, Csiszar A, Ungvari Z. Obesity-induced cognitive impairment in older adults: a microvascular perspective. Am J Physiol Heart Circ Physiol. 2021 Feb 1;320(2):H740-H761. doi: 10.1152/ajpheart.00736.2020. Epub 2020 Dec 18. PMID 33337961
- [Background] United Nations. (2019). World Population Prospects 2019: Highlights. UN. https://doi.org/10.18356/13bf5476-en
- [Background] Ferrucci L. The Baltimore Longitudinal Study of Aging (BLSA): a 50-year-long journey and plans for the future. J Gerontol A Biol Sci Med Sci. 2008 Dec;63(12):1416-9. doi: 10.1093/gerona/63.12.1416. No abstract available. PMID 19126858
- [Background] Tesfaye S, Cronin RM, Lopez-Class M, Chen Q, Foster CS, Gu CA, Guide A, Hiatt RA, Johnson AS, Joseph CLM, Khatri P, Lim S, Litwin TR, Munoz FA, Ramirez AH, Sansbury H, Schlundt DG, Viera EN, Dede-Yildirim E, Clark CR. Measuring social determinants of health in the All of Us Research Program. Sci Rep. 2024 Apr 16;14(1):8815. doi: 10.1038/s41598-024-57410-6. PMID 38627404
- [Background] Glynn NW, Santanasto AJ, Simonsick EM, Boudreau RM, Beach SR, Schulz R, Newman AB. The Pittsburgh Fatigability scale for older adults: development and validation. J Am Geriatr Soc. 2015 Jan;63(1):130-5. doi: 10.1111/jgs.13191. Epub 2014 Dec 31. PMID 25556993
- [Background] Ruderman SA, Webel AR, Willig AL, Drumright LN, Fitzpatrick AL, Odden MC, Cleveland JD, Burkholder G, Davey CH, Fleming J, Buford TW, Jones R, Nance RM, Whitney BM, Mixson LS, Hahn AW, Mayer KH, Greene M, Saag MS, Kamen C, Pandya C, Lober WB, Kitahata MM, Crane PK, Crane HM, Delaney JAC. Validity Properties of a Self-reported Modified Frailty Phenotype Among People With HIV in Clinical Care in the United States. J Assoc Nurses AIDS Care. 2023 Mar-Apr 01;34(2):158-170. doi: 10.1097/JNC.0000000000000389. Epub 2023 Jan 18. PMID 36652200
- [Background] Al Snih S, Chen NW, Chou LN, Markides KS, Ottenbacher KJ. Life Expectancy in Pre-Frail and Frail States with and without Disability: 18-Years of Follow-Up Data from the HEPESE Study Using the Markov Chain Method. J Frailty Aging. 2023;12(4):311-315. doi: 10.14283/jfa.2023.37. PMID 38008982
- [Background] D'Agostino RB Sr, Grundy S, Sullivan LM, Wilson P; CHD Risk Prediction Group. Validation of the Framingham coronary heart disease prediction scores: results of a multiple ethnic groups investigation. JAMA. 2001 Jul 11;286(2):180-7. doi: 10.1001/jama.286.2.180. PMID 11448281
- [Background] Casillas JM, Hannequin A, Besson D, Benaim S, Krawcow C, Laurent Y, Gremeaux V. Walking tests during the exercise training: specific use for the cardiac rehabilitation. Ann Phys Rehabil Med. 2013 Oct;56(7-8):561-75. doi: 10.1016/j.rehab.2013.09.003. Epub 2013 Sep 27. PMID 24126080
- [Background] . Lanting, S. (n.d.). Reliability and Validity of the PROMIS-57 Health Outcome Measures. ResearchGate. Retrieved October 28, 2024, from https://www.researchgate.net/publication/256326767_Reliability_and_Validity_of_the_PROMIS-57_Health_Outcome_Measures
- [Background] Hebert, K., Altidor, D., Tzoucalis, S., Mathews, A., & Dahl, W. (2023). Test-Retest Reliability of the MIND Diet Screener in Oldest-Old Adults. Journal of Nutrition Education and Behavior, 55(7, Supplement), 57-58. https://doi.org/10.1016/j.jneb.2023.05.128
- [Background] Young DR, Jee SH, Appel LJ. A comparison of the Yale Physical Activity Survey with other physical activity measures. Med Sci Sports Exerc. 2001 Jun;33(6):955-61. doi: 10.1097/00005768-200106000-00015. PMID 11404661
- [Background] Jiang L, Wang Y, Zhang Y, Li R, Wu H, Li C, Wu Y, Tao Q. The Reliability and Validity of the Center for Epidemiologic Studies Depression Scale (CES-D) for Chinese University Students. Front Psychiatry. 2019 May 21;10:315. doi: 10.3389/fpsyt.2019.00315. eCollection 2019. PMID 31178764
- [Background] Wechsler, D. (n.d.). Weschsler Adult Intelligence Scale: 4th Edition (WISC-IV) Pearson Assessments US. Retrieved October 28, 2024, from https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Wechsler-Adult-Intelligence-Scale-%7C-Fourth-Edition/p/100000392.html
- [Background] Wechsler, D. (n.d.). WAIS-IV Spain-Escala de inteligencia de Wechsler para adultos Cuarta edición, Spain Version Pearson Assessments US. Retrieved October 28, 2024, from https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Escala-de-inteligencia-de-Wechsler-para-adultos-%7C-Cuarta-edici%C3%B3n%2C-Spain-Version-/p/P100022001.html
- [Background] Wechsler, D. (n.d.). Escala de Memoria de Wechsler Cuarta Edición, Spain Version. Retrieved October 28, 2024, from https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Escala-de-Memoria-de-Wechsler-%7C-Cuarta-Edici%C3%B3n%2C-Spain-Version/p/P100038003.html
- [Background] Wechsler, D. (2009). Wechsler Memory Scale Fourth Edition. https://www.pearsonassessments.com/store/usassessments/en/Store/Professional-Assessments/Cognition-%26-Neuro/Wechsler-Memory-Scale-%7C-Fourth-Edition/p/100000281.html
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Northern Virginia Regional Commission. (n.d.). Demographics Northern Virginia Regional Commission-Website. Retrieved October 28, 2024, from https://www.novaregion.org/118/Demographics
- [Background] US Census Bureau. (n.d.). 2020 Census Results. Census.Gov. Retrieved October 28, 2024, from https://www.census.gov/2020results
- [Background] American College of Sports Medicine. (n.d.). Rankings. ACSM_CMS. Retrieved October 28, 2024, from https://www.acsm.org/about/community-impact-programs/american-fitness-index/rankings